CLINICAL TRIAL: NCT00362713
Title: A Phase 1b Safety and Dose-Assessment Study of Neoadjuvant Ipilimumab Monotherapy in Patients With Urothelial Carcinoma Undergoing Surgical Resection
Brief Title: Study of Neoadjuvant Ipilimumab in Patients With Urothelial Carcinoma Undergoing Surgical Resection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA184-027; NCT00462930 (obsolete NCT alias)
Record Dates: First submitted 2006-08-07; First posted 2006-08-10 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2009-12

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): 3 mg/kg or 10 mg/kg
  Interventions: Drug: Ipilimumab

INTERVENTIONS:
Drug: Ipilimumab — Intravenous Solution, Intravenous, One dose every 3 weeks for four weeks, followed through Week 24
  Other Names: BMS-734016; MDX-010

SUMMARY:
The purpose of this study is to learn if ipilimumab can be given safely at two different doses given to patients with urothelial cancer who are going to have surgery as part of their treatment. The immunological effectiveness of ipilimumab will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated urothelial cancer requiring surgery for treatment
* Ineligible for chemotherapy
* Adequate hematologic, kidney and liver function

Exclusion Criteria:

* Sexually active and fertile individuals or partners of these individuals who are unwilling or unable to use an acceptable method of birth control for the entire trial and up to 4 weeks after the study
* Women who are pregnant or breastfeeding
* Women with a positive pregnancy test on enrollment prior to study drug administration
* Prior treatment with ipilimumab or other anti-CTLA4 antibody, or a CD137 agonist
* Concurrent malignancy, with the exception of adequately treated and cured basal or squamous cell skin cancer, or carcinoma in situ of the cervix (previous malignancy without evidence of disease for 5 years will also be allowed to enter trial)
* Autoimmune disease: subjects with a documented history of inflammatory bowel disease (including Crohn's disease and ulcerative colitis) are excluded from this study as are patients with a history of symptomatic disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], Systemic Lupus Erythematosus, autoimmune vasculitis [e.g., Wegener's Granulomatosis]). Subjects with motor neuropathy considered of autoimmune origin (e.g., Guillain-Barre Syndrome) are excluded from this study
* Patients deemed ineligible for surgery
* Any non-oncology vaccine therapy used for prevention of infectious diseased in the past month
* Concomitant therapy with any of the following: IL-2, interferon or other non-study immunotherapy regimens, chemotherapy; immunosuppressive agents; other investigation therapies; or chronic use of systemic corticosteroids (used in the management of cancer or non-cancer related illnesses)
* Prior radiation therapy for urothelial cancer
* Positive screening tests for or any prior history of HIV, Hepatitis B or Hepatitis C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-03; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Safety of two dose levels of ipilimumab, given prior to surgery, in this patient population. | assessed throughout the study

SECONDARY OUTCOMES:
To evaluate anti-cancer immunological activity in blood and tissue samples compared to pre-treatment or control samples. | assessed throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- The University Of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx